CLINICAL TRIAL: NCT04591665
Title: Swallowing Changes in Cervical Spine Patients With Postoperative Dysphagia
Brief Title: Swallowing Difficult Sensation After Cervical Spine Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202008024RINC
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2020-10

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: swallowing examination — patients received swallowing examination, including high resolution impedance manometry and Video-Fluoroscopic swallowing study.

SUMMARY:
In many cases, the manometric examination is not feasible because of the pharyngeal sinusitis or pharyngeal torsion. In addition, although previous conventional manometry was used to estimate pharyngeal swallowing, the bolus flow transmission was still not evaluated, which still depended on the videofluoscopic swallowing studies. High resolution impedance manometry could help us to measure the bolus flow according to the impedance changes. However, the comparison between two approach methods of postoperative recovery of swallowing function is still inconclusive. The investigator aimed to examine the correlation between high-resolution manometric and videofluoroscopic measurements of the swallowing function.

DETAILED DESCRIPTION:
Background: In many cases, the manometric examination is not feasible because of the pharyngeal sinusitis or pharyngeal torsion. In addition, although previous conventional manometry was used to estimate pharyngeal swallowing, the bolus flow transmission was still not evaluated, which still depended on the videofluoscopic swallowing studies. High resolution impedance manometry could help us to measure the bolus flow according to the impedance changes. However, the comparison between two approach methods of postoperative recovery of swallowing function is still inconclusive.

Objectives: The objective of the current study was to examine the correlation between high-resolution manometric and videofluoroscopic measurements of the swallowing function.

Patients and methods: Consecutive patients who will fulfill the criteria of postoperative cervical spine surgery patients aged >= 20 will be enrolled and the dysphagia questionnaire score (EAT-10) was higher than 3, including 3. After got the inform consent, these patients receive the swallowing function by videofluroscopy and HRIM.

Expected result: The investigator will evaluate the swallowing changes of these postoperative cervical spine patients with suspected dysphagia. The investigator expected that the highly correlation between the HRIM and VFSS.

ELIGIBILITY:
Inclusion Criteria:

* > 20 years old
* postoperative cervical spine surgery
* EAT-10 questionnaire

Exclusion Criteria:

* pregnancy
* bleeding tendency
* heart or lung failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after cervical spine surgery, EAT-10 and older than 20 years old
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
pharyngeal pressure | 15 minutes
  the muscle power of pharyngeal contractility

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
ethical concern